CLINICAL TRIAL: NCT00943462
Title: Use of PET/CT Imaging With 18F-fluoroethylcholine (FEC) in the Evaluation of Patients Treated With Radiotherapy and Temozolomide Following a Diagnosis of Glioblastoma Multiforme
Brief Title: Study of 18F-FEC for Positron Emission Tomography-Computed Tomography (PET-CT) Imaging of GBM
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patients could be recruited.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Other Study IDs: CE-08-234; Schering-P06046
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Astrocytoma, Grade IV; Giant Cell Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glioblastoma Multiforme (GBM): We will conduct a prospective study on 20 consecutive patients who are seen at the Hôpital Notre-Dame neuro-oncology clinic for a diagnosis of GBM and who meet our inclusion criteria. We will meet with the eligible patients in order to provide them with a detailed description of the study procedures as well as to have them sign a consent form.
  Interventions: Radiation: External-beam radiation therapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: External-beam radiation therapy — 60 Gy of external beam radiotherapy using a standard technique will be administered in 2-Gy fractions, for a total of 30 fractions
Drug: Temozolomide — The chemotherapy will have to be administered in accordance with the protocol used in the CAN-NCIC-CE3 study, which established the current standard for treatment of GBM with the administration of temozolomide as adjuvant therapy at the same time as radiotherapy (clinicaltrials.gov ID NCT00006353).

SUMMARY:
Positron Emission Tomography-Computed Tomography (PET-CT) with injection of 18F-fluoroethylcholine (FEC) could be a useful tool in the evaluation and follow-up of patients who have been diagnosed with glioblastoma multiforme (GBM) and who are treated with radiotherapy and temozolomide by allowing, for example, the distinction of necrosis from tumour tissue. This tool could help the clinician in making therapeutic decisions for GBM patients.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 70 years of age
* Histological diagnosis of GBM (grade IV astrocytoma based on the World Health Organization [WHO] classification)
* No previous radiotherapy or chemotherapy
* No history of previous neoplasms
* Inoperable patients (tumour in place, biopsy only)
* KPS ≥ 70
* Adequate hematological, renal and hepatic function

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥ 100,000 per mm3
  * Serum creatinine ≤ 1.5 times the upper limit of normal of the laboratory where it is measured
  * Total bilirubin ≤ 1.5 times the upper limit of normal of the laboratory where it is measured
  * Liver enzymes < 3 times the upper limit of normal of the laboratory where they are measured
* Patients under corticosteroids must have received a stable or decreasing dose in the 14 days preceding randomization
* Consent form signed by the patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GBM patients seen at the neuro-oncology clinic of Centre hospitalier de l'Université de Montréal (CHUM)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Andrée Fortin, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)

REFERENCES:
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895